CLINICAL TRIAL: NCT01267435
Title: Study of Evaluation of Tibial and Femoral Tunnel Position After ACL Reconstruction
Brief Title: Evaluation of Tibial and Femoral Tunnel Position After Arthroscopic Reconstruction of the Anterior Cruciate Ligament
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Dr. Alireza Yousefy/Associate Professor of Medical Education, Shaheed Beheshty University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: ASD-1213-8
Record Dates: First submitted 2010-12-27; First posted 2010-12-28 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2008-10

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: Arthroscopy, Anterior Cruciate Ligament, Tibial Tunnel.
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- determining correct tunnel positions (Other)
  Interventions: Procedure: Anterior cruciate ligament reconstruction

INTERVENTIONS:
Procedure: Anterior cruciate ligament reconstruction — reconstruct the anterior cruciate ligament rupturing
  Other Names: ACL reconstruction

SUMMARY:
The purpose of this study is to evaluate the accuracy of tunnel positions in anterior cruciate ligament reconstruction

DETAILED DESCRIPTION:
The tunnel placement in ACL reconstruction is the most important predictor of clinical outcome and there is a high rate of inaccurate tunnel placements, even when performed by experienced surgeons.Tibial and femoral tunnel positions are one of the major concerns in anterior cruciate ligament reconstruction which have a great impact on the final surgical results

ELIGIBILITY:
Inclusion Criteria:

* anterior cruciate ligament rupturing

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
number of correct femoral tunnel position | 5 min after operation
  we evalauted femoral tunnel positions

SECONDARY OUTCOMES:
number of correct Tibial tunnel position | 5 min after operation
  we evalauted tibial tunnel position

CONTACTS AND LOCATIONS:
Overall Officials: hamidreza shemshaki, MD, Study Chair — research comittee
Locations (1):
- Akhtar university hospital, Tehran, Tehran Province, Iran